## Clinical Evaluation of Pneumatic Technology for Powered Mobility Devices

NCT03898362

July 3, 2025

Statistical Analysis Plan

Participants' demographics (e.g., age, gender, and race) were summarized using descriptive statistics. The phone interviews were recorded and then transcribed. During the focus group, the moderator took notes and summarized comments from Veterans and healthcare professionals. ATLAS.ti qualitative data analysis software was used to code and organize data from focus groups and interviews into themes. Overall, theme descriptions were influenced by the RESNA Wheelchair Service Provision Guide, which describes the "appropriate framework for identifying the essential steps in the provision of a wheelchair." The provision guide details the steps of the Provision Process: 1) referral, 2) assessment, 3) equipment recommendation and selection, 4) funding and procurement, 5) fitting, training and delivery, 6) follow-up, maintenance and repair, and 7) outcome measurements. The themes generated fit within one or more of these steps.